CLINICAL TRIAL: NCT05629416
Title: The Communicate Study Partnership - Improving Healthcare Experiences and Outcomes for Aboriginal Peoples Through Delivery of Culturally Safe Healthcare in First Languages
Brief Title: The Communicate Study Partnership
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Menzies School of Health Research (Other)
Collaborators: Northern Territory of Australia as represented by the Department of Health (Unknown); Djalkiri Foundation Aboriginal Corporation (Unknown); Charles Darwin University (Other); National Accreditation Authority for Translators and Interpreters (Unknown); Northern Territory Government as represented by the Department of The Chief Minister and Cabinet (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2008644
Record Dates: First submitted 2022-11-07; First posted 2022-11-29 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Aboriginal Health; Cultural Safety; Access to Interpreters; Healthcare Provider Training

STUDY DESIGN:
Intervention Model Description: Interventions to transform the culture of healthcare systems to achieve excellence in providing culturally safe care for First Nations peoples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cultural safety training and behaviour change intervention (Experimental): - Interventions to transform the culture of healthcare systems to achieve excellence in providing culturally safe care for First Nations peoples
  Interventions: Behavioral: Interventions to transform the culture of healthcare systems to achieve excellence in providing culturally safe care for First Nations peoples

INTERVENTIONS:
Behavioral: Interventions to transform the culture of healthcare systems to achieve excellence in providing culturally safe care for First Nations peoples — 1. Implement 'Ask the Specialist Plus', a structured program to promote anti-racism within Northern Territory (NT) hospitals by giving healthcare providers training in cultural safety.
  2. Implement strategies to foster 'Clinical champions of cultural safety' through a social media chat platform and face to face meetings to discuss anti-racism practice, cultural safety and practical ways to deliver culturally safe care including interpreter use.
  3. Support simplified and improved strategies for booking an interpreter to increase uptake.
  4. Implement retention strategies to ensure interpreters receive workplace support.
  5. Provide training in health terminology for interpreters.
  6. Integrate interpreter supply and demand through efficiency and effectiveness strategies tailored to participating sites.
  7. Implement continuous quality improvement cycles with senior managers, using findings from qualitative and quantitative data collection and evaluation.

SUMMARY:
The vision of the Communicate Study Partnership is to ensure more Aboriginal patients receive culturally safe healthcare in their first language.

The Communicate Study Partnership will implement and evaluate creative ways to embed cultural safety training and increase use of Aboriginal Interpreters and Aboriginal Health Practitioners at Northern Territory Top End hospitals.

Quantitative outcomes (interpreter uptake, outcomes including leave against medical advice, costs) will be measured using time-series analysis. Qualitative outcomes derived from interviews with patient, healthcare provider and interpreter participants, will be informed by decolonising theory and participatory approaches.

Successful project implementation will improve experience of care and health outcomes for Aboriginal people, build Aboriginal workforce, and improve healthcare provider satisfaction.

DETAILED DESCRIPTION:
The goal of "The Communicate Study: partnership across the Top End to improve Aboriginal patients' experience and outcomes of healthcare" is to achieve sustainable organisational change to provide excellence in cultural and clinical safety for Aboriginal people utilising NT Health facilities.

Aim 1: Transform the culture of healthcare systems to achieve excellence in providing culturally safe care for First Nations peoples

- Develop, implement and evaluate anti-racism training using 'Ask the specialist-Plus'. This comprises moderated discussion and reflection on 'Ask the Specialist' podcast episodes held during in-service and clinical teaching timeslots for healthcare providers

Aim 2: Strengthen the tools and strategies required underpinning culturally safe practice

1. Improve demand for Aboriginal interpreters and Aboriginal health practitioners through improved cultural understanding and recognition of patient needs
2. Improve supply of interpreters and Aboriginal health practitioners willing to work in the hospital environment by creating a culturally safe workplace and supporting career pathways
3. Effectiveness strategies tailored to participating sites such as

   * positioning interpreters at points of need and embedding them in medical and surgical teams
   * Optimising workflow to facilitate efficiency and availability across hospital departments

Aim 3: Evaluate outcomes using comprehensive qualitative and quantitative measures

1. Qualitative enquiry to assess cultural safety from patient perspectives, and understand experiences of Aboriginal and Non-Aboriginal healthcare providers and interpreters
2. Quantitative outcomes including

   * performance across key indicators: changes in documentation of language; Interpreter bookings made; Interpreter bookings completed; % Aboriginal patients in need getting access to an interpreter
   * Impact of intervention: proportion of admissions with and without interpreters ending in self-discharge; unplanned re-admissions and changes in hospital length of stay
   * economic analysis of the costs and cost benefits of interpreter use to decrease self-discharge and re-admission rates.

ELIGIBILITY:
Inclusion Criteria:

Different patient and provider participants (e.g. Aboriginal patients, Aboriginal interpreters, healthcare providers of any ethnicity) will be invited to participate in interviews, observations and surveys to assess effectiveness of study activities

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2022-05-23 (Actual); Primary Completion 2026-05-11 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Self discharge among Aboriginal inpatients at Royal Darwin Hospital, Palmerston Hospital, Katherine Hospital and Gove District Hospital | Up to 4 years. (Health system level data are collected and summarised quarterly during July 1 2022 - June 30 2026, and compared with the baseline phase July 1 2020 - June 30 2022)
  Self discharge (also referred to as 'Discharge against medical advice,', 'take own leave' or 'incomplete care') will be assessed among all admitted Aboriginal patients every quarter as a measure of the effeciveness of hospital-level study activities
  * Measured as proportion of all admissions of Aboriginal people that end in self-discharge
  * Data source: hospital Admitted Patient Care dataset (routinely collected by health services)
  The study has a two-year baseline phase July 1 2020 - June 30 2022, and four-year intervention (activity) period July 1 2022 - June 30 2026.
  There are no individually enrolled participants followed up at given time points; instead, activities are implemented continually at the level of the health systems, and outcomes are assessed using continuous hospital data and qualitative data, summarised quarterly.
Patient experience (qualitative evaluation) | Up to 4 years. Interview data will be collected at regular intervals throughout the study (2022-2026) to track any change in patient experience during the course of the intervention period
  Patient experience pre- and post-implementation of the interventions will be assessed through in-depth 30-60 minute one-on-one, face-to-face interviews of inpatients and patients who have recently (within 14 days) been discharged, by a member of the research team. The research team member will speak the patient's first language, or will work with an Aboriginal interpreter to conduct the interview.
  Some individuals with repeated contact with healthservices (such as renal dialysis patients) will be invited to participate in serial interviews over time

SECONDARY OUTCOMES:
Documentation of language in hospital medical records | Up to 4 years. (Documentation of language will be tracked throughout the 4-year intervention period.)
  Adequacy of documentation (proportion of Aboriginal patients for whom language is documented) will be used to inform quarterly quality improvement data review meetings. Data source: hospital electronic system (currently CARESYS, transitioning during the study period to ACACIA)
Access to an interpreter during admission | Up to 4 years. (Documentation of interpreter access will be tracked throughout the 4-year intervention period.)
  Interpreter access (proportion of Aboriginal patients with a language other than English as their first language) will be used to inform quarterly quality improvement data review meetings.
Healthcare provider experience | Up to 4 years. Interview data will be collected at regular intervals throughout the study (2022-2026) to track any change in healthcare provider experience during the course of the intervention period
  Healthcare provider experience of working with Aboriginal interpreters (qualitative evaluation) assessed by 30 minute semi-structured one-on-one, face-to-face interviews of healthcare providers with a member of the research team.
Cost | Up to 4 years. Continuous data (daily data, summarised monthly) will be assessed during - the two-year baseline phase July 1 2020 - June 30 2022 - the four-year intervention (activity) period July 1 2022 - June 30 2026
  Healthcare costs will be calculated based on variables including the top 6 ICD codes per admission and hospital length of stay. Economic evaluation will be conducted from the payer perspective and include the linked Admitted Patient Care and Aboriginal Interpreter Service datasets and NTHTE Unit expenditure reports, as well as ICD codes and Australian Refined DRGs.
Unplanned readmission within 28 days | Up to 4 years. Continuous data (daily data, summarised monthly) will be assessed during - the two-year baseline phase July 1 2020 - June 30 2022 - the four-year intervention (activity) period July 1 2022 - June 30 2026
  Continuous data collated monthly

CONTACTS AND LOCATIONS:
Overall Officials: Anna Ralph, PhD, Principal Investigator — Menzies School of Health Research
Locations (4):
- Australia (4):
  - Royal Darwin Hospital, Darwin, Northern Territory
  - Palmerston Hospital, Darwin, Northern Territory
  - Katherine Hospital, Katherine, Northern Territory
  - Gove District Hospital, Nhulunbuy, Northern Territory

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kerrigan V, McGrath SY, Herdman RM, Puruntatameri P, Lee B, Cass A, Ralph AP, Hefler M. Evaluation of 'Ask the Specialist': a cultural education podcast to inspire improved healthcare for Aboriginal peoples in Northern Australia. Health Sociol Rev. 2022 Jul;31(2):139-157. doi: 10.1080/14461242.2022.2055484. Epub 2022 Apr 3. PMID 35373706
- [Background] O'Connor E, Kerrigan V, Aitken R, Castillon C, Mithen V, Madrill G, Roman C, Ralph AP. Does improved interpreter uptake reduce self-discharge rates in hospitalised patients? A successful hospital intervention explained. PLoS One. 2021 Oct 12;16(10):e0257825. doi: 10.1371/journal.pone.0257825. eCollection 2021. PMID 34637434
- [Background] Kerrigan V, McGrath SY, Majoni SW, Walker M, Ahmat M, Lee B, Cass A, Hefler M, Ralph AP. "The talking bit of medicine, that's the most important bit": doctors and Aboriginal interpreters collaborate to transform culturally competent hospital care. Int J Equity Health. 2021 Jul 23;20(1):170. doi: 10.1186/s12939-021-01507-1. PMID 34301261
- [Background] Kerrigan V, McGrath SY, Majoni SW, Walker M, Ahmat M, Lee B, Cass A, Hefler M, Ralph AP. From "stuck" to satisfied: Aboriginal people's experience of culturally safe care with interpreters in a Northern Territory hospital. BMC Health Serv Res. 2021 Jun 4;21(1):548. doi: 10.1186/s12913-021-06564-4. PMID 34088326
- [Background] Mithen V, Kerrigan V, Dhurrkay G, Morgan T, Keilor N, Castillon C, Hefler M, Ralph AP. Aboriginal patient and interpreter perspectives on the delivery of culturally safe hospital-based care. Health Promot J Austr. 2021 Feb;32 Suppl 1:155-165. doi: 10.1002/hpja.415. Epub 2020 Dec 4. PMID 32888378
- [Background] Communicate Study group*. Improving communication with Aboriginal hospital inpatients: a quasi-experimental interventional study. Med J Aust. 2020 Aug;213(4):180-181. doi: 10.5694/mja2.50700. Epub 2020 Jul 25. No abstract available. PMID 32710454
- [Background] Kerrigan V, Lewis N, Cass A, Hefler M, Ralph AP. "How can I do more?" Cultural awareness training for hospital-based healthcare providers working with high Aboriginal caseload. BMC Med Educ. 2020 May 29;20(1):173. doi: 10.1186/s12909-020-02086-5. PMID 32471490
- [Background] Ralph AP, Lowell A, Murphy J, Dias T, Butler D, Spain B, Hughes JT, Campbell L, Bauert B, Salter C, Tune K, Cass A. Low uptake of Aboriginal interpreters in healthcare: exploration of current use in Australia's Northern Territory. BMC Health Serv Res. 2017 Nov 15;17(1):733. doi: 10.1186/s12913-017-2689-y. PMID 29141623
- See also: Project team's web page — https://www.menzies.edu.au/page/Research/Projects/Primary_health_care/The_Communicate_study/